CLINICAL TRIAL: NCT02725541
Title: Trial of Neoadjuvant Trastuzumab Emtansine in Patients With HER2-Equivocal Breast Cancer
Acronym: NATURE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: loss of funding support
Sponsor: Jenny C. Chang, MD (Other)
Collaborators: Genentech, Inc. (Industry); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Jenny C. Chang, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013875
Record Dates: First submitted 2016-03-18; First posted 2016-04-01 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: HER2 equivocal; Trastuzumab emtansine; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Trastuzumab emtansine at a dose of 3.6 mg/kg will be administered via intravenous infusion for 6 weeks (two 21-day cycles).
  Interventions: Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Trastuzumab emtansine — HER2-targeted antibody drug conjugate of trastuzumab and DM1
  Other Names: ado-trastuzumab emtansine; T-DM1; KADCYCLA

SUMMARY:
This is an open label, neoadjuvant phase II study to evaluate the objective response, toxicity, and safety of trastuzumab emtansine in patients with newly diagnosed HER2-equivocal breast cancer. Trastuzumab emtansine at a dose of 3.6 mg/kg will be intravenously administered every 3 weeks for a total of 6 weeks. Patients who achieve a partial or complete response after the 6-week treatment (responders) will continue on trastuzumab emtansine for an additional 12 weeks.

DETAILED DESCRIPTION:
NATURE is an open label, neoadjuvant, phase II study designed to evaluate the objective response rate of trastuzumab emtansine in patients with newly diagnosed HER2-equivocal breast cancer. Patients will receive trastuzumab emtansine at a dose of 3.6 mg/kg via intravenous infusion every 3 weeks for a total of 6 weeks (2 21-day cycles). Patients who achieve partial or complete response (responders) after the 6-week treatment will continue on trastuzumab emtansine for an additional 12 weeks (4 cycles). The primary objective will be objective response rate after 6 weeks of neoadjuvant trastuzumab emtansine. Secondary objectives will include imaging response (ultrasound and magnetic resonance imaging) after six weeks of neoadjuvant trastuzumab emtansine and toxicity and efficacy of trastuzumab emtansine. After completion of continued trastuzumab emtansine treatment, pathological complete response rate of responders as a whole and according to estrogen receptor status will be explored. Markers related to the mechanism of action of trastuzumab emtansine (HER2 copy number in circulating tumor cells; tissue expression of PTEN, PI3K, and other potential candidate markers) will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Female gender;
* Age ≥18 years;
* Eastern Cooperative Oncology Group performance status of 0-1;
* Histologically confirmed invasive breast cancer;
* Primary tumor greater than or equal to 1 cm diameter, as measured by clinical examination and mammography or ultrasound;
* Any N;
* No evidence of metastasis (M0) (isolated supra-clavicular node involvement allowed);
* HER2 low or equivocal status in the invasive component of the primary tumor (confirmed by a central certified laboratory prior to study entry)

  * HER2 low expression: 1+/2+ by immunohistochemistry and/or HER2/CEP17 ratio <2.0 with HER2 copy number <6.0 signals/cell
  * HER2 equivocal expression: HER2 copy number ≥4.0 and <6.0 signals/cell;
* Hematopoietic status:

Absolute neutrophil count ≥ 1.0 x 10^9/L, Platelet count ≥ 100 x 10^9/L, Hemoglobin at least 9 g/dL;

• Hepatic status: Serum total bilirubin ≤1 x upper limit of normal (ULN; In the case of known Gilbert's syndrome, a higher serum total bilirubin [< 1.5 x ULN] is allowed), Aspartate aminotransferase and alanine aminotransferase ≤1.5 x ULN, Alkaline phosphatase ≤ 1.5 x ULN;

• Renal status: Creatinine ≤1.5 mg/dL;

* International Normalized Ratio ≤1.5 x ULN;
* Baseline left ventricular ejection fraction ≥50%, as measured by echocardiography or multigated acquisition scan;
* Negative serum or urine β-human chorionic gonadotropin pregnancy test within 7 days prior study entry for patients of childbearing potential. Women of childbearing potential must use effective contraception (barrier method [condoms, diaphragm] in conjunction with spermicidal jelly, or total abstinence. Oral, injectable, and implantable hormonal contraceptives are not allowed) for the duration of the study and for at least 7 months after the last dose of study treatment;
* Signed informed consent form (ICF);
* Patient accepts to make available tumor samples for submission to central laboratory to conduct translational studies as part of this protocol.

Exclusion Criteria:

* Previous (less than 5 years) or current history of malignant neoplasms, except for curatively treated basal and squamous cell carcinoma of the skin and carcinoma in situ of the cervix;
* Patients with a prior malignancy diagnosed more than 5 years prior to study entry;
* Preexisting peripheral neuropathy ≥ grade 2;
* Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension (≥180/110), unstable diabetes mellitus, dyspnea at rest, or chronic oxygen therapy;
* Concurrent disease or condition that would make the patient inappropriate for study participation or any serious medical disorder that would interfere with the patient's safety;
* Unresolved or unstable serious adverse events from prior administration of another investigational drug;
* Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of ICF;
* Concurrent neoadjuvant cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy other than the trial therapy);
* Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trastuzumab emtansine or its components;
* Ejection fraction <55% or below the lower limit of the institutional normal range;
* Pregnant or lactating women;
* Concomitant use of cytochrome P450 3A4 inhibitors or inducers;
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol;
* Active infection requiring intravenous or oral antibiotics;
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 weeks
  Determine the objective response rate after 6 weeks of neoadjuvant trastuzumab emtansine (RECIST 1.1)

SECONDARY OUTCOMES:
Radiological response | 6 weeks
  Determine radiological response after 6 weeks of neoadjuvant trastuzumab emtansine
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 18 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03

OTHER OUTCOMES:
Pathological complete response (pCR) rate | 18 weeks
  Determine the pCR rate of continued trastuzumab emtansine treatment in responders
pCR rate | 18 weeks
  Determine the pCR rate of continued trastuzumab emtansine treatment in responders according to estrogen receptor status
Correlative markers of trastuzumab emtansine response | 6 weeks
  Explore correlative markers of trastuzumab emtansine response using tumor biopsy specimens

CONTACTS AND LOCATIONS:
Overall Officials: Jenny C. Chang, M.D., Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and materials on human subjects will be shared with other eligible investigators through appropriate means in accordance with the NIH policy on Sharing Research Data (NIH Guide, February 26, 2003). Data will be also shared with the funding agency and regulatory agencies as required. Data will be shared with other investigators within the limits of HIPAA and other patient confidentiality requirements. This will generally require removal of all patient identifiers for all source documents and the use of arbitrarily assigned one-way identifiers. In some cases, requestors will be asked to sign a formal data sharing agreement that will provide for a commitment to use data only for research purposes and not to identify individuals, keep the data secure, and destroy or return data after analyses are complete. Prior approval will be obtained from collaborating investigators, research sponsors, and/or other stake-holders before sharing if proprietary information or products are involved.